CLINICAL TRIAL: NCT02668146
Title: A Double-Blind, Cross-Over, Placebo-Controlled Efficacy and Tolerability Study of Perampanel and Essential Tremor
Brief Title: An Efficacy/Safety Study of Perampanel for Reducing Essential Tremor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Adrian Handforth, MD, Assistant Chief of Staff, Neurology VAGLAHS, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0042
Record Dates: First submitted 2015-10-28; First posted 2016-01-29 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Essential Tremor
Keywords: essential tremor; Perampanel; clinical trial
MeSH Terms: conditions — Essential Tremor | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- perampanel (Experimental): Perampanel administration
  Interventions: Drug: Perampanel
- placebo (Placebo Comparator): Placebo administered to subjects.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Perampanel — Study drug will be administered to study subjects
  Arms: perampanel
Drug: Placebo — Placebo will be administered to study subjects
  Arms: placebo

SUMMARY:
Obtain information on whether the medication Perampanel reduces tremor in people with essential tremor and is well-tolerated.

DETAILED DESCRIPTION:
Please see descriptions in "Primary and Secondary Outcomes".

ELIGIBILITY:
Inclusion Criteria:

1. Subject has reviewed, signed and dated a written informed consent form and use of protected health information [Health Insurance Portability and Accountability Act (HIPAA) Authorization], including videotaping consent.
2. Subject is 18 or older.
3. Subject has a diagnosis of definite or probable essential tremor (ET) as defined by the Tremor Investigational Group, with involvement of the hands and arms of at least 2 years duration, without present causes of enhanced physiologic tremor, no recent exposure to tremorogenic drugs or drug withdrawal states, no direct or indirect trauma to the nervous system within 3 months preceding the onset of tremor, and no historic or clinical evidence of psychogenic tremor origin.
4. Tremor severity score of at least 2 in at least one upper extremity on the Fahn-Tolosa-Marin Tremor Rating Scale, or at least 1.5 on the TETRAS scale.
5. Subject is taking the same dose of one to three anti-tremor medications for at least 4 weeks prior to screening, has an inadequate response to that/those medication(s), and, barring any unforeseen circumstances, will continue for the duration of the study on the same dose(s) of anti-tremor medication(s), OR Has failed at least one course of an anti-tremor medication and cannot tolerate available anti-tremor medication(s), OR Is naive to anti-tremor treatment and refuses to take available anti-tremor medications.
6. If a woman of childbearing potential:

   A. Must be unable to become pregnant or use adequate birth control; B. Must be defined as status post hysterectomy or tubal ligation, or 2 years post-menopausal, OR C. Otherwise documented to be incapable of pregnancy, or have practiced one of the following methods of contraception for at least two months prior to screening: 1) hormonal contraceptives, 2) spermicide and barrier method, 3) intrauterine device, 4) partner sterility, 5) abstinence, and have a negative pregnancy test during screening.
7. Subject is accessible by telephone.
8. Subject can comply with study visits, study drug compliance, and study procedures.
9. Subject is on stable doses of all other medications for at least 4 weeks prior to the first baseline visit, and, barring any unforeseen circumstances, for the duration of the study

   -

Exclusion Criteria:

1. Subject's tremor is adequately controlled on a current treatment.
2. Subject is pregnant, plans to become pregnant during the study or within 2 months of completing the study or who is presently lactating or breast-feeding.
3. Subject has other medical conditions that may cause or explain subject's tremor, such as but not limited to, Parkinson's disease, hyperthyroidism, pheochromocytoma, head trauma or cerebrovascular disease within 3 months prior to the onset of essential tremor; multiple sclerosis, polyneuropathy or family history of Fragile X syndrome.
4. Subject taking medication(s) that might produce tremor or interfere with the evaluation of tremor, such as but not limited to: CNS-stimulants, stimulant decongestants, beta-agonist bronchodilators, lithium, amiodarone, metoclopramide, theophylline, valproate, Irregular use ("as needed" or "prn") of benzodiazepines, sleep medications or anxiolytics; (However, regular use of a benzodiazepine, sleep medication or anxiolytic to improve sleep or performance is allowed as long as tremor persists against the background of regular medication use)
5. Subject has had surgical intervention for their tremor in the past (e.g., ablative thalamotomy or gamma knife thalamotomy), or has had a botulinum toxin injection in the 6 months prior to screening
6. Subject has used an experimental drug within the 4 weeks prior to screening (or within 5 half-lives, whichever is longer) for any reason, OR has used a device for the treatment of essential tremor in the 4 weeks prior to screening, OR has ever used deep brain stimulation for any reason
7. Subject cannot abstain from the use of the following drugs for the stated period of time prior to a clinic visit: caffeine (8 hours) and alcohol (12 hours).
8. Subject cannot abstain from use of alcohol prior to driving vehicle or operating heavy machinery.
9. Subject with a history in the last 2 years of alcohol or substance abuse (DSM 305); or history of consuming more than 2 glasses of wine (or equivalent) per day in the last 28 days prior to screening.
10. Subject with a history of significant psychiatric disorder (e.g., mania, bipolar depressive disorder, schizophrenia, schizoaffective disorder, or other major psychiatric disorder), significant coagulation, immunologic, gastrointestinal, respiratory, cardiovascular (e.g., uncontrolled hypertension, myocardial infarction in the last 18 months, significant bundle branch block, congestive heart disease), endocrine (e.g., uncontrolled diabetes, hyperthyroidism) disorder, or current or chronic infection, significant Screening laboratory or ECG abnormalities, or any acute or chronic illness or abnormality which in the opinion of the Investigator precludes study participation. Subject with Right Bundle Branch Block, pacemakers, controlled asthma or controlled hypertension and/or controlled diabetes (hemoglobin A1c < 8%) are acceptable, as are subjects with thyroid disease, provided they are euthyroid on treatment. Subject with single or recurrent episodes of major depressive disorder (DSM IV 296.20 -.25 or 296.30-.35) that have been successfully managed with a stable dose (over 60 days) of an antidepressant may be considered for entry.
11. Subject with liver disease that is more than mild. This is defined as transaminase levels AST and ALT greater than 50% above normal.
12. Subject with severe renal disease, defined as having creatinine clearance less than 39 ml/min.
13. Subject has had a suicide attempt, suicidal ideation with intent, or history of aggression, including but not restricted to violence or threat of violence, within the past 2 years.
14. Subject with a recent history of hematologic/oncologic disorders (within 2 years), other than successfully resolved cutaneous basal cell or squamous cell carcinomas. Stability after treatment for prostate cancer is also acceptable.
15. Subject with clinically significant impaired balance or considered at increased risk for falls.
16. Subject is taking phenytoin, carbamazepine, oxycarbazine, rifampin, St John's wart, ketonazole or consuming grapefruit juice.
17. Subject with history of taking perampanel in the past. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Tremor reduction. TETRAS scale, performance sub scale. | 40 weeks
  This scale evaluates tremor of various body parts during postures, movement and tasks. Items are scored from 0 to 4, with 4 representing highest severity. Maximum score is 64.
Tremor reduction. TETRAS scale. Activity of Daily Living subscale. | 40 weeks
  The subject rates to what extent tremor affects activities in a 12-item, 0-to-4 scale. Maximum score is 48.
Tremor reduction. TETRAS scale. Subject Global Impression of Change. | 40 weeks
  Subjects rate the degree of change from minus 3 to plus 3.
Tremor reduction. TETRAS scale. QUEST subscale (QUality of life in Essential Tremor). | 40 weeks
  30-item questionnaire in which the subject rates on a 0 to 4 scale how much tremor affects aspects of life.
Safety. vitals; | 40 weeks
  Weight (lbs), respiration rate (rps), heart rate (bps) and blood pressure (mmhg).
Tolerability. Adverse Events. | 40 weeks
  At each clinic and phone visit, the PI and coordinator will collect information on any adverse events. An Adverse Event will be defined as any clinically undesirable event.
Safety; laboratory testing | 40 weeks
  At each clinic visit. Laboratory testing will be done. This will include metabolic panel (serum electrolytes, glucose (mg/dl) , creatinine (mg/dl) , calcium (mg/dl), magnesium (mg/dl), Complete Blood Count(CBC) (mg/dl), White Blood Count (WBC) (k/ul), platelets (k/ul), hepatic panel (total BILIRUBIN, Total PROTEIN, ALKALINE PHOSPHATASE, ALANINE AMINOTRANSFERASE, ASPARTATE AMINOTRANSFERASE, ALBUMIN GLUTAMYL TRANSFERASE LDH), and urinalysis.
Safety. Laboratory testing; screen visit testing | screen visit
  Screen Visit testing will include hemoglobin A1c (%), free thyroxin (ng/dl), and Thyroid Stimulating Hormone (TSH) (uIU/mL) . An EKG will be performed.

SECONDARY OUTCOMES:
Treatment effects on Daily Living (The QUEST scale to assess quality of life) | 40 weeks
  Assess the effect of treatment on tremor-affected activities of daily living. The QUEST scale to assess quality of life in essential tremor. It is a 30-item questionnaire in which the subject rates on a 0 to 4 scale how much tremor affects aspects of life
QOLIE changes | 40 weeks
  Assess changes in Quality Of Life (QOLIE).
Subjective assessment of global life changes | 40 weeks
  Assess subject global impression of change as a result of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Charles A Handforth, M.D., Principal Investigator — VHAGLAHS
Locations (1):
- VA Greater Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No